CLINICAL TRIAL: NCT05677802
Title: Examining the Feasibility of Implementing a Biobehavioral Stress Reduction Program in Triple Negative Breast Cancer Patients
Brief Title: Feasibility Study of Biobehavioral Stress Reduction Intervention in Patients With Triple Negative Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Samilia Obeng-Gyasi, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: OSU-22083; NCI-2022-08781 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-12-15; First posted 2023-01-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; HER2-Negative Breast Carcinoma; Hormone Receptor-Negative Breast Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health Services Research (stress management therapy) (Experimental): Patients receive biobehavioral stress reduction intervention while on study. Patients undergo blood specimen collection at baseline and follow up and have their medical records reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Medical Chart Review; Procedure: Stress Management Therapy; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Medical Chart Review — Undergo medical cart review
  Other Names: Chart Review
Procedure: Stress Management Therapy — Receive biobehavioral stress reduction intervention
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial aims to see if patients with triple negative breast cancer can complete a biobehavioral stress reduction program that also addresses health related social needs (e.g., utilities, transportation, etc.). The stress reduction program is over ten weeks and includes stress reduction (e.g., progressive muscle relaxation), coping, problem solving, communication, and social support. Health related social needs will be evaluated at the beginning of the study, and referrals will be made to social work to help address those needs. The study will examine stress as reported by the patients and also use biological markers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I Acceptability of the biobehavioral intervention will be determined using the Client Satisfaction Questionnaire (CSQ). CSQ is an 8-item self-report measure with item assessing different aspects of treatment satisfaction (e.g., quality of service, the degree to which needs were met, overall satisfaction).

III Tolerability of the biobehavioral intervention will be assessed by analyzing pre to post treatment change on the Profile of Mood States.

III Feasibility of the biobehavioral intervention will be assessed using three metrics: 1) accrual number as a percentage of available patients approached; 2) number/percent of patients completing each BBI session; and, 3) number/percent of patients retained and completing 10 BBI sessions.

SECONDARY OBJECTIVE:

I. To examine the feasibility of collecting biomarkers--white blood cell count, C-reactive protein, Interleukin-6, TNF-alpha (α), systolic blood pressure, diastolic blood pressure, heart rate, total cholesterol, high-density lipoprotein; albumin, hemoglobin A1C, body mass index (BMI).

EXPLORATORY OBJECTIVE:

I. To test for pre/post effects of the biobehavioral stress reduction intervention on measures of stress (Impact of Events Scale), mood and psychological symptoms, and allostatic load.

OUTLINE:

Patients receive biobehavioral stress reduction intervention while on study. Patients undergo blood specimen collection at baseline and follow up, and have their medical records reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Untreated newly diagnosed triple negative breast cancer
* Stages I-III

Exclusion Criteria:

* Prisoners
* Male
* Identifying as American Indian, Alaska Native, Asian, Native Hawaiian or Other Pacific Islander
* Individuals not able to speak and understand English
* Known personal history of ductal carcinoma in situ (DCIS) or invasive breast cancer
* Stage IV breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Participant Satisfaction with the Biobehavioral Intervention | Up to 2 years
  Acceptability will be measured at the end of the intervention using the Client Satisfaction Questionnaire (CSQ). CSQ scores range from 8-32 with higher scores indicating higher satisfaction.
Profile of Mood States for the Biobehavioral Intervention | Up to 2 years
  This will be assessed analyzing pre to post treatment change on the Profile of Mood States short form. The Profile of Mood States short from is a 37 item survey with lower scores indicative of stable mood.
Participant Biobehavioral Intervention | Up to 2 years
  Feasibility will be evaluated using three metrics: 1) accrual number as a percentage of available patients approached; 2) number/percent of patients completing each Biobehavioral intervention (BBI) session; and, 3) number/percent of patients retained and completing 10 BBI sessions.

SECONDARY OUTCOMES:
Biomarkers for allostatic load | Up to 2 years
  The points for each biomarker will be summarized into a total score ranging from 0-12. The pre-test allostatic load biomarker will be based on the distribution of each biomarker within the study sample at diagnosis. For each biomarker, each patient will be stratified into quartiles. A point will be assigned for membership in the worst quartile. The post-test allostatic load will be calculated similar to the pre-test allostatic load using biomarkers collected after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Samilia Obeng-Gyasi, MD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - MetroHealth, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu